CLINICAL TRIAL: NCT03970278
Title: A Long-Term Follow-up Study to Evaluate the Safety and Efficacy of Adeno Associated Virus (AAV) Serotype 8 (AAV8)-Mediated Gene Transfer of Glucose-6-Phosphatase (G6Pase) in Adults with Glycogen Storage Disease Type Ia (GSDIa)
Brief Title: Study of Long-Term Safety and Efficacy on Gene Therapy in Glycogen Storage Disease Type Ia
Status: Completed | Type: Observational
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: 401GSDIA02; 2018-004473-27 (EudraCT Number); 2023-504004-29-00 (EU CTIS Number)
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Glycogen Storage Disease Type IA; Von Gierke's Disease (GSD Type Ia)
Keywords: AAV; gene therapy; glucose metabolism disorder; carbohydrate metabolism, inborn errors; genetic diseases; Inborn Metabolic Diseases
MeSH Terms: conditions — Hepatorenal form of glycogen storage disease; Glycogen Storage Disease Type I; Glucose Metabolism Disorders; Carbohydrate Metabolism, Inborn Errors; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | US Export: No

GROUPS / COHORTS (1):
- All Participants: All participants enrolled in study 401GSDIA02 will have received a single IV dose of DTX401(pariglasgene brecaparvovec) during their participation in study 401GSDIA01 (NCT03517085).
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The primary objective of this study is to determine the long-term safety of DTX401 following a single intravenous (IV) dose in adults with GSDIa.

DETAILED DESCRIPTION:
Only participants who received DTX401 in study 401GSDIA01 (NCT03517085) are eligible to participate in study 401GSDIA02. No investigational product will be administered during study 401GSDIA02.

ELIGIBILITY:
Inclusion Criteria:

1. Received DTX401 in study 401GSDIA01.
2. Willing and able to provide written informed consent after the nature of the study has been explained, and prior to any research-related procedures being performed.
3. Willing and able to comply with all scheduled study visits, procedures, and requirements.

Exclusion Criteria:

1. Planned or current participation in any other interventional clinical study that may confound the safety or efficacy evaluation of DTX401 during this study.
2. Presence or history of any condition that, in the view of the Investigator, poses a risk to subject safety or places the subject at high risk of poor compliance or not completing the study or that would significantly affect the interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects 18 years of age or older with GSDIa previously enrolled in 401GSDIA01.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs), Serious AEs and Discontinuations Due to AEs | Up to 312 weeks following DTX401 administration

SECONDARY OUTCOMES:
Change in Time to First Hypoglycemic Event During a Controlled Fasting Challenge from Day 0 (Study 401GSDIA01) to 312 weeks | Up to 312 weeks following DTX401 administration

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (6):
- United States (3):
  - UCONN Health, Farmington, Connecticut
  - Michigan Medicine University of Michigan, Ann Arbor, Michigan
  - University of Texas Health Science Center at Houston, Houston, Texas
- Montreal Children Hospital, McGill University Health Centre, Montreal, Quebec, Canada
- University Medical Center Groningen, Groningen, Netherlands
- Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, A Coruna, Spain

IPD SHARING:
Plan to Share IPD: No
Due to the rarity of GSDIa and the small number of subjects in this trial, individual patient data will not be shared in order to safeguard patient privacy, consistent with the data sharing commitment statement listed on Ultragenyx.com.